CLINICAL TRIAL: NCT01635335
Title: A Randomized Controlled Trial of Family-Based HIV Prevention for Latino Youth
Brief Title: Randomized Control Trial of Family-Based HIV Prevention for Latinos
Acronym: LatinoSTYLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Celia Lescano, Research Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01MH087232 (NIH); 5R01MH087232 (NIH)
Record Dates: First submitted 2012-06-30; First posted 2012-07-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: HIV; Sexually Transmitted Infections
Keywords: HIV prevention; adolescents; Latinos; Hispanics; family; health promotion; disease prevention; family communication; parental supervision
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV-specific (Experimental): 7-hour multiple family workshop focused on providing information and skills related to HIV prevention. Specific focus on parent-adolescent communication and parental monitoring.
  Interventions: Behavioral: Latino STYLE
- General Health Promotion (Active Comparator): 7-hour multiple family workshop focused on providing information related to various adolescent health risk behaviors, including smoking, alcohol, violence, nutrition, and exercise.
  Interventions: Behavioral: Latino STYLE

INTERVENTIONS:
Behavioral: Latino STYLE — 7-hour family-based workshop with 3-hour follow-up booster 3 months later

SUMMARY:
The proposed project will test an HIV prevention intervention for Latino parent-adolescents dyads. This randomized controlled trial will:

1. Recruit and randomize 320 parent-adolescent dyads into a Latino family-based HIV prevention intervention or a family-based General Health Promotion condition.
2. Determine the efficacy of the Latino Family-based HIV prevention intervention from assessment of changes in HIV-related sexual behavior and attitudes over 18 months among a sample of 320 Latino parent-adolescent dyads.
3. Determine the efficacy of the Latino Family-based HIV prevention intervention from assessment of changes in family relationships and parental monitoring/supervision over 18 months among a sample of 320 Latino parent-adolescent dyads.
4. Examine the association of other important constructs, such as religiosity, acculturation, cultural values, and sexual socialization with the primary outcomes.

Based on a thorough review of the literature and preliminary data from a recent, small pilot study, the investigators hypotheses are:

1. Compared to the General Health Promotion Control condition, the Family-Based HIV Prevention intervention will result in greater change with regard to primary outcome measures of safer sexual behavior (recent sexual activity, the number of unprotected sex acts, and intentions to use condoms) and safer HIV-related attitudes.
2. Compared to the General Health Promotion Control condition, the Family-Based HIV Prevention intervention will result in greater change with regard to family relationships and parental monitoring/supervision through improved parent-child communication skills and they will mediate the intervention impact.
3. Religiosity, acculturation, cultural values, and sexual socialization will have meaningful associations with the primary outcomes and will act as moderators of intervention impact.

DETAILED DESCRIPTION:
Latinos are disproportionately represented among those diagnosed with HIV and Latino adolescents are at risk for engaging in sexual behaviors that can lead to HIV. To date, data regarding HIV prevention interventions for Latino adolescents, as distinct from other ethnic groups, have been rare. Thus, an efficacious HIV prevention intervention is urgently needed for Latino adolescents. The current proposal is aimed at filling that gap by evaluating a newly developed family-based intervention that incorporates cultural constructs into the Social-Personal Framework.

This R01 builds on the Principal Investigator's NIMH-funded K Award, which piloted a culturally-specific family-based intervention with 80 Latino parent-adolescent dyads and demonstrates promising results. Extending this work, 320 Latino parent-adolescent dyads with an adolescent between the ages of 14 and 17 will be randomized into either the family based HIV prevention intervention or a family-based general health promotion control condition. In both conditions, the interventions will use a multi-family group format consisting of 6 to 8 parent and youth dyads in a one-day, 7-hour workshop. Both interventions employ activities for youth and parents separately (e.g., focus on adolescent vulnerability) and parents and adolescents together (e.g., address parent/adolescent communication). The project will determine the efficacy of the Latino Family-based HIV prevention intervention from assessment of changes in the adolescents' HIV-related sexual behavior and attitudes, gender and sexual socialization, parent-child communication, and parental monitoring. Measures will be completed at baseline and at 3, 6, 12, and 18 months post-intervention.

HIV/AIDS is a significant problem in the Latino community. Developing culturally sensitive HIV prevention interventions for Latino youth, in particular, is a public health priority. Family-based interventions are likely to be well received by the Latino population. Therefore, this project will examine the efficacy of a family-based HIV prevention intervention for Latino youth and parents to decrease the incidence of HIV among Latinos. Its innovation is in being one of the first to work with Latinos specifically in a family-based intervention where parents and adolescents come together to discuss important sexuality-related topics.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and parents self-identify as Latino/Hispanic
* Adolescents between the ages of 14 and 17
* Parent is Spanish-Speaking and feels comfortable speaking Spanish in groups
* Adolescent is English-speaking and feels comfortable speaking English in groups
* Adolescent meets behavioral inclusion criteria (not disclosed)

Exclusion Criteria:

* Adolescent self-discloses HIV positive status
* Currently or intending to be pregnant during the course of the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2010-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in sexual activity status | baseline and 3, 6, 12, and 18 months post-intervention

SECONDARY OUTCOMES:
Change in Unprotected Sex Acts | baseline and 3, 6, 12, and 18 months post-intervention
  change in the number of incidences of unprotected vaginal or anal intercourse
Change in intentions to use condoms | baseline and 3, 6, 12, and 18 months post-intervention
Change in parent-adolescent communication | baseline and 3, 6, 12, and 18 months post-intervention
change in parental monitoring of adolescent | baseline and 3, 6, 12, and 18 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Celia Lescano, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Lescano CM, Castillo HL, Calcano E, Mayor M, Porter M, Rivera-Torgerson Y, Dion C, Marhefka SL, Barker D, Brown LK; Latino STYLE Research Group. Latino STYLE: Preliminary Findings From an HIV Prevention RCT Among Latino Youth. J Pediatr Psychol. 2020 May 1;45(4):411-422. doi: 10.1093/jpepsy/jsaa019. PMID 32330945
- See also: related info — http://www.facebook.com/projectlatinoSTYLE